CLINICAL TRIAL: NCT02158507
Title: An Open Label, Pilot Study of Veliparib (ABT-888) and Lapatinib (Tykerb) in Patients With Metastatic, Triple Negative (ER, PR, and HER-2 Negative) Breast Cancer
Brief Title: Pilot Study of Veliparib (ABT-888) and Lapatinib (Tykerb) in Patients With Metastatic, Triple Negative Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Breast Cancer Research Foundation of Alabama (Unknown); GlaxoSmithKline (Industry); AbbVie (Industry)
Responsible Party: Principal Investigator, Erica Stringer-Reasor, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F131219003 (UAB 1372); 000504723 (Other: Office of Sponsored Programs)
Record Dates: First submitted 2014-05-29; First posted 2014-06-09 (Estimated); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Triple Negative Breast Cancer
Keywords: triple negative breast cancer (TNBC); Veliparib; Lapatinib; estrogen receptor negative; progesterone receptor negative; (HER-2-Neu) negative
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Lapatinib; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination of Veliparib + Lapatinib (Experimental): Lapatinib will be administered as a tablet at a dosage of 1250 mg/day continuously for 28 days starting on Day 1 of each cycle. Veliparib will be administered as a capsule at a dosage of 200 mg every 12 hours for 28 days starting on Day 2 of each cycle. A cycle of therapy is defined as 28 days. Treatment is administered on an outpatient basis. Patient response will be evaluated every 8 weeks according to the current Response Evaluation Criteria in Solid Tumors (RECIST) guidelines and performance of relevant scans and/or x-rays.
  Interventions: Drug: Combination of Veliparib + Lapatinib

INTERVENTIONS:
Drug: Combination of Veliparib + Lapatinib — Treatment cannot be in administered conjunction with other chemotherapy, targeted therapy, radiation therapy, or other investigational drugs.
  Other Names: Veliparib (ABT-888); Lapatinib (Tykerb)

SUMMARY:
This study will evaluate the effectiveness and safety of the combination of two drugs, Veliparib and Lapatinib, given to participants with metastatic triple negative breast cancer that have undergone previous treatment. Veliparib is an investigational drug and has not been approved by the FDA while Lapatinib has been approved by the FDA for another type of breast cancer. All eligible participants will receive the study medications and not a placebo.

DETAILED DESCRIPTION:
Breast cancer is the most commonly diagnosed cancer in American women. Metastatic breast cancer remains incurable partially due to the lack of targeted therapy for selected subsets of patients. There are five distinct subsets of breast cancer with unique biological profiles. Triple negative breast cancer (TNBC) is a subset with special clinical interest because of its significant percentage of occurrence (10-20% of all breast cancer diagnoses) and its poor prognosis. With no defined targeted therapy to date, this study seeks to investigate a therapeutic strategy based on specific molecular abnormalities in the tumor cells of TNBC.

ELIGIBILITY:
Inclusion Criteria:

* Patient must pathologically documented stage IV breast cancer.
* Tumor must be HER-2 negative, and estrogen and progesterone receptors negative. Patients with BRCA 1 or 2 mutations will not be included.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension.
* Biopsy of a metastatic lesion is not required for protocol entry but all patients with reasonably accessible lesions must agree to biopsy. (Lung and brain metastasis will not be biopsied.) Patients with no reasonably accessible lesions can be enrolled in the trial.
* Prior Therapy:

  * No more than two regimens in the metastatic setting as long as patients have adequate performance status. Patients with no prior chemotherapy for metastatic disease may be included in the trial if they received anthracyclines and taxanes in the adjuvant or neoadjuvant settings. Chemotherapy naïve patients with metastatic disease must have failed anthracyclines and taxanes.
  * Chemotherapy treatment prior to enrollment must be discontinued for at least 3 weeks prior to study entry.
  * Patients must have completed radiation therapy at least 21 days prior to beginning protocol treatment.
* Patients must have recovered from all reversible toxicities related to prior therapy before beginning protocol treatment and may not have an pre- existing treatment-related toxicities higher than Grade 2. Patients must have less than Grade 2 pre-existing peripheral neuropathy.
* Patients may receive bisphosphonates. However, if used, bone lesions may not be used for progression or response.
* At least 19 years of age.
* Life expectancy of >12 weeks.
* Performance status according to Eastern Cooperative Oncology Group (ECOG) is less than or equal to 2.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count: greater than or equal to 1,000/uL
  * Hemoglobin: greater than or equal to 9 mg/dL
  * Platelets: greater than or equal to 100,000/uL
  * Total bilirubin: less than or equal to 1.5 times the institutional upper limit of normal
  * AST (SGOT)/ALT (SGPT): less than or equal to 2.5 times the institutional upper limit of normal without liver metastases OR less than or equal to 5 times the institutional upper limit of normal if documented liver metastases
  * Creatinine: less than or equal to 1.5 mg/dL OR calculated creatinine clearance greater than or equal to 40 mL/min (calculated using the modified Cockcroft and Gault method).
* Ability to understand and the willingness to sign a written informed consent document.
* Use of an effective means of contraception in subjects of child-bearing potential.
* Negative serum or urine beta-HCG (human chorionic gonadotropin) pregnancy test at screening for patients with childbearing potential.
* Ejection fraction must be 50%.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* No prior use of anthracyclines and taxanes for metastatic disease or in the adjuvant or neoadjuvant setting.
* Metastatic lesions identifiable only by PET.
* QTc (corrected QT) >470 msec. Excluded are patients who may develop prolongation of QTc. These conditions include patients with hypokalemia or hypomagnesemia, congenital long QT syndrome, patients taking anti- arrhythmic medicines or other medicinal products that lead to QT prolongation, and cumulative high-dose anthracycline therapy.
* Patients may not be receiving concurrent chemotherapy for treatment of metastatic disease.
* Active brain metastases: evidence of progression less than or equal to 3 months after local therapy. (Patients should be asymptomatic and off corticosteroids and anticonvulsants for at least 3 months prior to study entry).
* Patients with brain metastases must have at least one site of measurable disease outside of the central nervous system.
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, history of recent myocardial infarction, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease or psychiatric illness/social situations that would limit compliance with study requirements.
* Uncontrolled seizure disorder.
* Pregnant or lactating women are excluded. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated. These potential risks may also apply to other agents used in this study.
* A prior invasive malignant disease within five years except for skin cancer (squamous cell or basal cell carcinoma).
* Patients with known history of HIV or Hepatitis B because of potential for added toxicity from treatment regimen.
* Dementia or altered mental status that would prohibit the understanding of informed consent.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andres Forero, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stringer-Reasor EM, May JE, Olariu E, Caterinicchia V, Li Y, Chen D, Della Manna DL, Rocque GB, Vaklavas C, Falkson CI, Nabell LM, Acosta EP, Forero-Torres A, Yang ES. An open-label, pilot study of veliparib and lapatinib in patients with metastatic, triple-negative breast cancer. Breast Cancer Res. 2021 Mar 4;23(1):30. doi: 10.1186/s13058-021-01408-9. PMID 33663560
- See also: An open-label, pilot study of veliparib and lapatinib in patients with metastatic, triple-negative breast cancer | Breast Cancer Research — https://link.springer.com/article/10.1186/s13058-021-01408-9#Sec22

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination of Veliparib + Lapatinib
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combination of Veliparib + Lapatinib
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 50 [37 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing Study-related Toxicities When Taking Veliparib in Combination With Lapatinib
Description: Drug related toxicities for the safety analysis are defined as: a) any grade 3 or 4 non-hematologic toxicity except alopecia and nausea which is not refractory to anti-emetics; b) failure to recover to baseline (except alopecia) after delaying the next dose by more than 14 days; c) grade 3 or 4 neutropenia complicated by fever equal to or greater than 38.50 degrees C or infection, or grade 4 neutropenia of a least 7 days duration; or d) grade 4 thrombocytopenia, or grade 3 thrombocytopenia complicated by hemorrhage. Toxicity evaluation of the patients enrolled in the trial will be done using the NCI Common Toxicity Criteria.
Time Frame: baseline to 4 years
Measure: Number; unit: count of participants
Arm/Group | Combination of Veliparib + Lapatinib
Number analyzed (Participants) | 17
count of participants
  fatigue | 6
  diarrhea | 5
  constipation | 5
  insomnia | 5
  vomiting | 3
  anemia | 3
  headache | 3
  dizziness | 2
  dyspnea | 2
  rash | 2

2. Secondary Outcome: Number of Subjects With Objective Response Rate (ORR) at 4 Years Post Baseline (Complete Responses [CRs] Plus Partial Responses [PRs]
Description: Complete responses plus partial responses will be included as indicators of an objective response rates. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 4 years post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Combination of Veliparib + Lapatinib
Number analyzed (Participants) | 17
Participants | 17

3. Secondary Outcome: Number of Subjects With Progression Free Survival (PFS) at 4 Years After Start of Study.
Description: Number of subjects who survive to 4 years with no disease progression. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Baseline to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Combination of Veliparib + Lapatinib
Number analyzed (Participants) | 17
Participants | 17

4. Secondary Outcome: DNA Methylation and RNA Transcriptome Will be Evaluated Before and After Therapy; Baseline Pattern Will be Compared With the Post Treatment Pattern to Identify Markers of Response or Resistance.
Description: Analysis of the genomic data from tumors may allow us to identify if there is a gene or groups of genes that will be able to predict response or resistance to the research combination; in order to conduct the genomic evaluation it is necessary to correlate with clinical response. In addition, we will conduct IHC studies in order to analyze markers that will indicate us if the combination of the research agents inhibit the targets for which they were designed (H2AX, BRCA and EGFR); this data needs to be correlated with clinical data to see if the lab evaluations correlate with the response of the patient. In addition, we will evaluate by IHC markers of apoptosis that will indicate us if the combination of research agents was cytotoxic against the tumor cells ; this data needs to be correlated with clinical data to see if the lab evaluations correlate with the response of the patient.
Time Frame: Within 4 weeks of baseline (treatment initiation)
Population: Progressive Disease (PD)/Partial Response (PR)=Fold Change
Measure: Number; unit: percentage of fold change
Arm/Group | Combination of Veliparib + Lapatinib
Number analyzed (Participants) | 17
percentage of fold change
  CALML5 | -15.74
  MMP7 | -12.45
  BRCA1 | -4.82
  PLA2G3 | 4.74
  CRYAB | -4.55
  COL11A1 | -4.48
  CKB | -4.36
  LFNG | 4.13
  RASGRF1 | -3.79
  PIK3R3 | -3.6
  SOCS1 | 3.46
  GJB2 | 3.15
  PTCH1 | -3.05
  STAT1 | 2.96
  COL27A1 | -2.57
  SOCS2 | 2.53
  FGFR2 | -2.49
  NOTCH1 | -2.27
  HGF | 2.21

5. Secondary Outcome: Measure Numbers of Circulating Tumor Cells Before and After Therapy
Description: Circulating tumor cells will be measured before and after therapy and will indicate if the therapy is active against the tumor; a decrease in the number of the circulating tumor cells will indicate effectiveness of the combination.
Time Frame: Before and after Cycle 1 (up to 28 days)
Population: This lab test was not performed. Circulating Tumor Cells were no longer clinically relevant upon IRB approval of this study. This was inadvertently not removed from the protocol or CT.gov outcome measures at the start of the study.
  CTC was being studied by a different investigator (Dr. Haluska) was at Mayo at the initial writing of the protocol and subsequently left and was never with UAB
Measure: Number; unit: participants
Arm/Group | Combination of Veliparib + Lapatinib
Number analyzed (Participants) | 0

6. Secondary Outcome: Peak Plasma Concentration of Veliparib and Palatinib When Given in Combination.
Description: Blood samples for the first day will be collected 5 minutes before the start of therapy, 30 and 60 minutes after the first dose of Lapatinib and then 2, 4, 6, 8, and 24 hours after the start of Lapatinib. On day 2, Lapatinib and Veliparib will be given and samples will be taken 30 and 60 minutes after the first dose and then at 2, 4, 6, 8, and 24 hours. Additional blood samples will be taken on day 3, before the third day dose of the combined study drugs. The same schema will be followed on days 8, 9, and 10.
  Each pharmacokinetic variable will be divided by dose groups for descriptive statistical analyses (mean, standard deviation, coefficient of variation, geometric mean, median, minimum and maximum per dose group).
Time Frame: Up to day 10
Measure: Median (Full Range); unit: nanograms per mL
Arm/Group | Combination of Veliparib + Lapatinib
Number analyzed (Participants) | 17
nanograms per mL | 2600 [2300 to 2900]

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Combination of Veliparib + Lapatinib
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 17/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination of Veliparib + Lapatinib (N=17)
fatigue (Nervous system disorders) | 17 (17)
diarrhea (Gastrointestinal disorders) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT02158507/Prot_SAP_000.pdf